CLINICAL TRIAL: NCT01370902
Title: A Randomised, Double-blind, Placebo-controlled, Single-dose and Multiple-dose, Dose-escalation Trial Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0141-0000-0100 in Subjects With Rheumatoid Arthritis
Brief Title: Safety and Tolerability of NNC0141-0000-0100 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8765-3658; 2010-019234-28 (EudraCT Number); U1111-1120-2542 (Other: WHO)
Record Dates: First submitted 2011-05-31; First posted 2011-06-10 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single-dose (SD) trial part (i.v.) (Experimental)
  Interventions: Drug: NNC 0141-0000-0100; Drug: placebo
- Single-dose (SD) trial part (s.c.) (Experimental)
  Interventions: Drug: NNC 0141-0000-0100; Drug: placebo
- Multiple-dose (MD) trial part (s.c.) (Experimental)
  Interventions: Drug: NNC 0141-0000-0100; Drug: placebo

INTERVENTIONS:
Drug: NNC 0141-0000-0100 — Single dose administered subcutaneously (under the skin), up to six dose levels. Progression to next dose will be based on safety evaluation. Initiation of the MD s.c. phase will depend on the results from the SD i.v. cohorts as well as the first two dose cohorts of the SD s.c. part
  Arms: Single-dose (SD) trial part (s.c.)
Drug: placebo — Single dose administered subcutaneously (under the skin) as a comparator at all dose levels
  Arms: Single-dose (SD) trial part (s.c.)
Drug: NNC 0141-0000-0100 — Multiple doses administered subcutaneously (under the skin) at 4 different occasions with a dosing interval of two weeks, at five different dose levels.
  Arms: Multiple-dose (MD) trial part (s.c.)
Drug: placebo — Multiple doses administered subcutaneously (under the skin) as a comparator at all dose levels
  Arms: Multiple-dose (MD) trial part (s.c.)
Drug: NNC 0141-0000-0100 — Single dose administered intravenously (into a vein), up to nine dose levels. Progression to next dose will be based on safety evaluation. Initiation of the SD s.c. phase will depend on the results from the first three dose cohorts of the SD i.v. part
  Arms: Single-dose (SD) trial part (i.v.)
Drug: placebo — Single dose administered intravenously (into a vein), as a comparator at all dose levels
  Arms: Single-dose (SD) trial part (i.v.)

SUMMARY:
This trial is conducted in Europe. The aim of this dose-escalating trial is to assess the safety, tolerability, pharmacokinetics (the rate at which the body eliminates the trial drug) and pharmacodynamics (the effect of the investigated drug on the body) of single and repeated doses of NNC141-0100 in subjects with Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of rheumatoid arthritis (RA) according to the American College of Rheumatology (ACR1987 classification) of at least 3 months duration prior to randomisation
* Active Rheumatoid Arthritis (RA) characterised by a DAS28-CRP (Disease Activity Score of 28 joints, calculated with CRP (C-reactive protein) value) greater than or equal to 3.2
* Females must be post-menopausal or surgically sterile (post-menopausal for at least 1 year) or be willing to use highly effective method of birth control
* Males must be willing to use highly effective contraception
* Subjects on stable doses of methotrexate (7.5 to 25 mg/week, both inclusive) for at least 4 weeks prior to randomisation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | from trial product administration to week 12

SECONDARY OUTCOMES:
Antibodies against NNC141-0100 | from trial product administration until final visit (week 12 or longer if applicable)
Area under the serum concentration-time curve - SD trial part | from trial product administration until final visit (week 12 or longer if applicable)
Terminal half-life (t½) - SD trial part | from trial product administration until final visit (week 12 or longer if applicable)
Terminal half-life (t½) - MD trial part | from trial product administration until final visit (week 12 or longer if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Buffet, Study Director — Innate Pharma
Locations (1):
- Berlin, Germany